CLINICAL TRIAL: NCT05408143
Title: An Enhanced Home-Based Telemedicine Program Using Remote Examination Devices for Children With Medical Complexity Receiving Comprehensive Care: a Single-Center Randomized Controlled Trial
Brief Title: An Enhanced Home-Based Telemedicine Program Using Remote Examination Devices for Children With Medical Complexity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Children and Youth with Special Health Care Needs National Research Network (CYSHC) (Unknown)
Responsible Party: Principal Investigator, Ricardo A. Mosquera, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-21-0829; 5 UA6MC31101-05-00 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2022-04-20; First posted 2022-06-07 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Chronic Diseases in Children
Keywords: Comprehensive Care; Telemedicine enhanced with TytoCare devices.; Telemedicine; children with medical complexity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- usual CC (with conventional telemedicine) (Active Comparator)
  Interventions: Other: CC
- comprehensive care (CC) augmented with enhanced telemedicine (ETM) (Experimental)
  Interventions: Other: CC; Device: enhanced telemedicine (ETM)

INTERVENTIONS:
Other: CC — To promote prompt effective care for medically complex children at all hours, we developed an outpatient comprehensive care (CC) program at the University of Texas Health Science Center at Houston (UTH) that now includes a hospital consultation service by the outpatient CC providers (the hospital component) and a conventional telemedicine (CTM) audio-visual program (the home component).
Device: enhanced telemedicine (ETM) — An enhanced telemedicine program (using HIPAA-compliant, mobile TytoCareTM devices) will be added to CC to allow providers to remotely visualize the skin, throat, & ears, auscultate the heart & lungs, and measure illnesses during clinic hours and chronic illnesses during the detailed patient evaluation to be conducted at least every 6 months by "virtual patient rounds" in the home. These visits will involve the parent(s), the PCP, and if needed any of 10 specialists, particularly pulmonology, gastroenterology, neurology, and physical medicine and rehabilitation. A social worker, nutritionist, or psychologist will be involved as needed. Each PCP will perform 2-3 virtual patient rounds per week to proactively identify medical problems, suboptimal adherence to treatment, dosing errors, or other problems and intervene before CMC develop a serious illness or require avoidable clinic visits, Emergency Department visits, or hospitalizations.
  Arms: comprehensive care (CC) augmented with enhanced telemedicine (ETM)

SUMMARY:
The purpose of this study is to assess if the benefits for children with medical complexity (CMC) receiving comprehensive care (CC) in an enhanced medical home can be further improved by enhanced telemedicine program (ETM) provided during clinic hours using mobile devices to measure temperature& oxygen saturation, auscultate the heart & lungs, and view the skin, throat, & tympanic membranes in the home.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 2 hospitalizations or greater than or equal to 1 ICU admission in the year before joining the comprehensive care program
* Greater than 50 percent estimated risk of hospitalization without our care as judged by the medical director

Exclusion Criteria:

* Major heart disease
* Mitochondrial disorders
* Active cancer
* Do-Not-Resuscitate (DNR) order
* Patients receiving compassionate care

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of days care provided in a medical setting | end of study(about 24 months)
Total number of episodes of serious illnesses (causing death, pediatric ICU admission, and hospital stay > 7d). | end of study(about 24 months)

SECONDARY OUTCOMES:
Cost effectiveness of ETM | end of study(about 24 months)
  this is defined strictly as a reduction in serious illnesses without an increase in health system costs, a decrease in health system costs without an increase in serious illnesses, or a reduction in both
All cause infections on admission to the hospital | end of study(about 24 months)
Total numbers of clinic visits | end of study(about 24 months)
Total number of emergency department visits | end of study(about 24 months)
Total number of hospital days | end of study(about 24 months)
Total number of Pediatric Intensive Care Unit (PICU) days | end of study(about 24 months)
Total number of deaths | end of study(about 24 months)
Parent ratings of care assessed using the Consumer Assessment of Healthcare Providers and Systems Survey | end of study(about 24 months)
  This survey consists of 5 questions. The first 4 are scored from 1(never)-4(always) for a maximum score of 16 , a higher number indicating better care. The fifth question is scored form 0-10 a higher number indicating a better provider.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Mosquera, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No